CLINICAL TRIAL: NCT00003804
Title: Nephroblastoma Clinical Trial and Study
Brief Title: Chemotherapy Plus Surgery in Treating Children at Risk of or With Stage I Wilms' Tumor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066948; SIOP-93-01; EU-98064
Record Dates: First submitted 1999-11-01; First posted 2004-07-16 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2012-04

CONDITIONS: Kidney Cancer
Keywords: stage I Wilms tumor
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — Dactinomycin; Vincristine

INTERVENTIONS:
Biological: dactinomycin
Drug: vincristine sulfate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known which regimen of chemotherapy is more effective for stage I Wilms' tumor.

PURPOSE: Randomized phase III trial to study the effectiveness of chemotherapy and surgery in treating children who are at risk of or who have stage I Wilms' tumor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the initial extension of disease, surgical procedures, gross and histological morphology, treatments, clinical outcome, and late consequences of therapy after treatment with neoadjuvant chemotherapy, surgery, and adjuvant chemotherapy with or without maintenance chemotherapy in patients with intermediate risk or anaplastic stage I Wilms' tumor. II. Determine the safety and effectiveness of reduced chemotherapy in these patients.

OUTLINE: This is a randomized, multicenter study. Patients receive dactinomycin IV on days 1-3 and 15-17 and vincristine IV on days 1, 8, 15, and 22. Patients then undergo surgery about a week after completion of chemotherapy. After surgery, patients receive vincristine IV on days 1, 8, 15, and 22 and dactinomycin IV on days 8-12. Patients are then randomized to one of two treatment arms after week 9. Arm I: Patients receive dactinomycin IV on days 1-5 of week 10 and vincristine IV on day 1 of both weeks 10 and 11. This course is repeated during weeks 17 and 18. Arm II: Patients receive no further treatment. Patients are followed every 3 months for 3 years, then annually thereafter. Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 350 patients (175 per treatment arm) will be accrued for this study within 7-8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Initial diagnosis of a unilateral tumor with clinical and radiological characteristics of a nephroblastoma Histologically proven stage I Wilms' tumor after neoadjuvant treatment and surgery Intermediate risk or anaplastic No detectable distant metastases 4 weeks after adjuvant chemotherapy

PATIENT CHARACTERISTICS: Age: 0.5 to 17 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 1993-07

CONTACTS AND LOCATIONS:
Overall Officials: Jan DeKraker, MD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (44):
- Clinique de l'Esperance, Montegnée, Belgium
- Clinical Hospital Center Split, Split, Croatia
- University Children Hospital, Brno, Czechia
- Denmark (3):
  - Aalborg Hospital, Aalborg
  - Universtiy Hospital of Aarhus, Aarhus
  - Odense University Hospital, Odense
- France (17):
  - Hopital Nord Amiens, Amiens
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - CHU de Bordeaux - Hopital Pellegrin, Bordeaux
  - C.H.U. de Brest, Brest
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Regional de Lille, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Hopital d'Enfants de la Timone, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHR Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - C.H.U. Saint Etienne Hospital Nord, Saint-Etienne
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier Regional de Purpan, Toulouse
  - C.H. Bastien de Clocheville, Tours
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Children's Hospital A. Kyriakou, Athens, Greece
- Ospedale Raffaele Silvestrini, San Sisto Perugia, Italy
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Emma Kinderziekenhuis, Amsterdam
  - University Medical Center Nijmegen, Nijmegen
- Norway (3):
  - Haukeland Hospital - University of Bergen, Bergen
  - University of Tromso, Tromsø
  - Regionsykehuset & University Hospital, Trondheim
- Wroclaw Medical University, Wroclaw (Breslau), Poland
- Hospital Escolar San Joao, Porto, Portugal
- Pediatricna Klinika, Ljubljana, Slovenia
- Spain (6):
  - Hospital General Universitari Vall d'Hebron, Barcelona
  - Centro Medico "La Zarzuela", Madrid
  - Hospital Universitario LaPaz, Madrid
  - Hospital Materno-Infantil, Málaga
  - Hospital General de Galicia, Santiago de Compostela
  - Hospital Des Cruces, Vizcaya
- Sweden (2):
  - Lund University Hospital, Lund
  - Karolinska Hospital, Stockholm
- Tawam Hospital, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] Sudour H, Audry G, Schleimacher G, Patte C, Dussart S, Bergeron C. Bilateral Wilms tumors (WT) treated with the SIOP 93 protocol in France: epidemiological survey and patient outcome. Pediatr Blood Cancer. 2012 Jul 15;59(1):57-61. doi: 10.1002/pbc.24059. Epub 2012 Jan 11. PMID 22238153
- [Background] Warmann SW, Nourkami N, Fruhwald M, Leuschner I, Schenk JP, Fuchs J, Graf N. Primary lung metastases in pediatric malignant non-Wilms renal tumors: data from SIOP 93-01/GPOH and SIOP 2001/GPOH. Klin Padiatr. 2012 Apr;224(3):148-52. doi: 10.1055/s-0032-1304600. Epub 2012 Apr 18. PMID 22513793
- [Background] Furtwangler R, Nourkami N, Alkassar M, von Schweinitz D, Schenk JP, Rube C, Siemer S, Leuschner I, Graf N. Update on relapses in unilateral nephroblastoma registered in 3 consecutive SIOP/GPOH studies - a report from the GPOH-nephroblastoma study group. Klin Padiatr. 2011 May;223(3):113-9. doi: 10.1055/s-0031-1275293. Epub 2011 Apr 20. PMID 21509706
- [Background] van den Heuvel-Eibrink MM, van Tinteren H, Rehorst H, Coulombe A, Patte C, de Camargo B, de Kraker J, Leuschner I, Lugtenberg R, Pritchard-Jones K, Sandstedt B, Spreafico F, Graf N, Vujanic GM. Malignant rhabdoid tumours of the kidney (MRTKs), registered on recent SIOP protocols from 1993 to 2005: a report of the SIOP renal tumour study group. Pediatr Blood Cancer. 2011 May;56(5):733-7. doi: 10.1002/pbc.22922. Epub 2010 Dec 22. PMID 21370404
- [Background] Warmann SW, Furtwangler R, Blumenstock G, Armeanu S, Nourkami N, Leuschner I, Schenk JP, Graf N, Fuchs J. Tumor biology influences the prognosis of nephroblastoma patients with primary pulmonary metastases: results from SIOP 93-01/GPOH and SIOP 2001/GPOH. Ann Surg. 2011 Jul;254(1):155-62. doi: 10.1097/SLA.0b013e318222015e. PMID 21670612
- [Background] van den Heuvel-Eibrink MM, Grundy P, Graf N, Pritchard-Jones K, Bergeron C, Patte C, van Tinteren H, Rey A, Langford C, Anderson JR, de Kraker J. Characteristics and survival of 750 children diagnosed with a renal tumor in the first seven months of life: A collaborative study by the SIOP/GPOH/SFOP, NWTSG, and UKCCSG Wilms tumor study groups. Pediatr Blood Cancer. 2008 Jun;50(6):1130-4. doi: 10.1002/pbc.21389. PMID 18095319
- [Background] Luithle T, Szavay P, Furtwangler R, Graf N, Fuchs J; SIOP/GPOH Study Group. Treatment of cystic nephroma and cystic partially differentiated nephroblastoma--a report from the SIOP/GPOH study group. J Urol. 2007 Jan;177(1):294-6. doi: 10.1016/j.juro.2006.09.011. PMID 17162067
- [Background] Szavay P, Luithle T, Graf N, Furtwangler R, Fuchs J. Primary hepatic metastases in nephroblastoma--a report of the SIOP/GPOH Study. J Pediatr Surg. 2006 Jan;41(1):168-72; discussion 168-72. doi: 10.1016/j.jpedsurg.2005.10.021. PMID 16410128
- [Result] Boccon-Gibod LA. Pathological evaluation of renal tumors in children: international society of pediatric oncology approach. Pediatr Dev Pathol. 1998 May-Jun;1(3):243-8. doi: 10.1007/s100249900033. PMID 10463285
- [Result] Fuchs J, Kienecker K, Furtwangler R, Warmann SW, Burger D, Thurhoff JW, Hager J, Graf N. Surgical aspects in the treatment of patients with unilateral wilms tumor: a report from the SIOP 93-01/German Society of Pediatric Oncology and Hematology. Ann Surg. 2009 Apr;249(4):666-71. doi: 10.1097/SLA.0b013e31819ed92b. PMID 19300220
- [Result] Furtwangler R, Reinhard H, Beier R, et al.: Clear-cell sarcoma (CCSK) of the kidney - results of the SIOP 93-01/GPOH trial. [Abstract] Pediatr Blood Cancer 45 (4 Suppl 1): A-0.155, 423, 2005.
- [Result] Ora I, van Tinteren H, Bergeron C, de Kraker J; SIOP Nephroblastoma Study Committee. Progression of localised Wilms' tumour during preoperative chemotherapy is an independent prognostic factor: a report from the SIOP 93-01 nephroblastoma trial and study. Eur J Cancer. 2007 Jan;43(1):131-6. doi: 10.1016/j.ejca.2006.08.033. Epub 2006 Nov 2. PMID 17084075
- [Result] Reinhard H, Aliani S, Ruebe C, Stockle M, Leuschner I, Graf N. Wilms' tumor in adults: results of the Society of Pediatric Oncology (SIOP) 93-01/Society for Pediatric Oncology and Hematology (GPOH) Study. J Clin Oncol. 2004 Nov 15;22(22):4500-6. doi: 10.1200/JCO.2004.12.099. PMID 15542800
- [Result] Reinhard H, Semler O, Burger D, Bode U, Flentje M, Gobel U, Gutjahr P, Leuschner I, Maass E, Niggli F, Scheel-Walter HG, Stockle M, Thuroff JW, Troger J, Weirich A, von Schweinitz D, Zoubek A, Graf N. Results of the SIOP 93-01/GPOH trial and study for the treatment of patients with unilateral nonmetastatic Wilms Tumor. Klin Padiatr. 2004 May-Jun;216(3):132-40. doi: 10.1055/s-2004-822625. PMID 15175957
- [Result] Verschuur AC, Vujanic GM, Van Tinteren H, Jones KP, de Kraker J, Sandstedt B. Stromal and epithelial predominant Wilms tumours have an excellent outcome: the SIOP 93 01 experience. Pediatr Blood Cancer. 2010 Aug;55(2):233-8. doi: 10.1002/pbc.22496. PMID 20582946
- [Result] Vujanic GM, Harms D, Bohoslavsky R, Leuschner I, de Kraker J, Sandstedt B. Nonviable tumor tissue should not upstage Wilms' tumor from stage I to stage II: a report from the SIOP 93-01 nephroblastoma trial and study. Pediatr Dev Pathol. 2009 Mar-Apr;12(2):111-5. doi: 10.2350/08-03-0432.1. Epub 2008 Sep 23. PMID 18811224